CLINICAL TRIAL: NCT04947345
Title: The Availability and Safety Study of Remimazolam Besylate for Injection on Sedation of ERAS Patients Under Mechanical Ventilation in ICU: Protocol for a Randomized, Open-label, Controlled Trial
Brief Title: The Availability and Safety Study of Remimazolam Besylate for Injection on Sedation of ERAS Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Yichang Humanwell Pharmaceutical Co., Ltd., China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-JS-2814
Record Dates: First submitted 2021-06-14; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Analgesia; Postoperative Pain
Keywords: sedative; Remimazolam Besylate; postoperative sedation
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Propofol

STUDY DESIGN:
Masking Description: This is a open label clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group: Remimazolam Besylate (Experimental): Patients should be given study drugs as soon as possible after entering the ICU. Syringe pump is used to administer medication. Loading dose of Remimazolam is 0.2 mg/kg, which is administered for less than 1 min initially. Maintaining dose is 0.2-1 mg/kg/h. Sedative target is RASS between 0 and -2 points. Excepts for fentanyl and Remimazolam, no analgesic or sedative could be used during the experimental time period.
  Interventions: Drug: Remimazolam Besylate
- Positive control group: Propofol (Active Comparator): Patients should be given study drugs as soon as possible after entering the ICU. Syringe pump is used to administer medication. Loading dose of propofol is 0.2 mg/kg, which is administered for less than 1 min initially. Maintaining dose is 0.3-4.0 mg/kg/h. Sedative target is RASS between 0 and -2 points. Excepts for fentanyl and propofol, no analgesic or sedative could be used during the experimental time period.
  Rescue therapy for experimental group During the treatment of the experimental group, if the RASS cannot be maintained at 0 to -2 points at the maximum Remimazolam maintenance dose of 1 mg/kg/h, a loading dose of propofol (0.2 mg/kg) can be given intravenously. If RASS fails to satisfied after three loading doses of propofol, Remimazolam is discarded and 0.3-4.0 mg/kg/h of propofol are used as rescue therapy for experimental group.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam Besylate — Remimazolam Besylate are used as sedatives for subjects in this arm.
  Arms: Experimental group: Remimazolam Besylate
Drug: Propofol — Propofol are used as sedatives for subjects in this arm.
  Arms: Positive control group: Propofol

SUMMARY:
This trial intends to evaluate Remimazolam Besylate's availability and safety compared with propofol.

ELIGIBILITY:
Inclusion criteria

* Meet criteria of enhanced recovery after surgery (ERAS);
* Mechanical ventilated when enrolled and have estimation of more than 10 hours of mechanical ventilation in ICU
* Aged between 18-75 years old AND 18kg/m2 ≤ BMI ≤ 30 kg/m2;
* Clearly know the purpose and objective of this clinical study and voluntarily enrolled.

Criteria of ERAS: (1) without dysfunction of nervous system or Glasgow Coma Score > 12; (2) a satisfied glucose level (random blood glucose<11.1mmol/L during screening stage) for diabetes mellitus patients; (3) Without acute coronary syndrome in recent 6 months; (4) Without bradycardia and third-degree atrioventricular block (except for patients with pacemaker) during screening stage; (5) systolic blood pressure>90mmHg with no usage of vasoactive agent during screening stage; (6) without mental illness (schizophrenia, depressive disorder), cognitive dysfunction (identified by MMSE), epilepsy, history of abuse of psychotropic or anesthesia medication; (7) without disorder of coagulation function (PT/INR/APTT > 1.5×upper limit), bleeding tendency (active peptic ulcer), under treatment of thrombolysis and anticoagulant; (8) without disorder of liver function (ALT/AST > 2×upper limit and total bilirubin>1.5×upper limit); (9) without disorder of renal function (Creatine or BUN/Urea>1.5×upper limit); without dialysis patients.

Exclusion criteria

* Allergy to component of Remimazolam besylate for injection;
* Woman in gestation and lactation period;
* Enrolled in other clinical trails in recent 3 months;
* Other circumstance that identified by researchers that do not suitable for this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Satisfaction rate of sedation | 24 hours since injection of sedatives
  (number of subjects that meets satisfied RASS score under prescribed dose of sedative agents during study / total number of subjects) ×100%
Rate of major clinical events | 48 hours since injection of sedatives
  (number of subjects that suffer from major clinical events during study / total number of subjects) ×100%. Major clinical events are defined as cardiac arrest, malignant arrhythmia, new onset of shock, new onset of sepsis and respirate failure unrelated to primary illness.

SECONDARY OUTCOMES:
incidence of delirium | 48 hours since injection of sedatives
  (subjects with delirium / total number of subjects ×100%) by 12h and 24h after entering ICU
Time to weaning and extubation | 48 hours since injection of sedatives
  Time to weaning and extubation
Difficulty of nursing | 48 hours since injection of sedatives
  By Barthel index assessment
28-days survival | 28 days since injection of sedatives
  (number of subjects that alive in 28-days since ICU entry/ total number of subjects) ×100%
incidence of rescue therapy in experimental group | 24 hours since injection of sedatives
  (number of subjects that receive rescue therapy in experimental group/ total number of subjects) ×100%

IPD SHARING:
Plan to Share IPD: Undecided
So far, we haven't decide if individual participant data are suitable to share with other researchers.

REFERENCES:
- [Derived] Liu S, Su L, Zhang B, He H, Li Z, Li Q, Wang Q, Smith F, Long Y. The Availability and Safety Study of Remimazolam Besylate for Injection on Sedation of ERAS Patients Under Mechanical Ventilation in ICU: Protocol for a Randomized, Open-Label, Controlled Trial. Front Med (Lausanne). 2021 Nov 5;8:735473. doi: 10.3389/fmed.2021.735473. eCollection 2021. PMID 34805204